CLINICAL TRIAL: NCT01654783
Title: Observational Study on Clinical Practice in the Management of Ulcerative Colitis With Oral 5-Aminosalicylic Acid in Japan
Brief Title: Observational Study in the Management of Ulcerative Colitis With Oral 5-ASA
Status: Completed | Type: Observational
Sponsor: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTIMUM-2012
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Ulcerative Colitis
Keywords: 5-ASA, ulcerative colitis, active, remission, adherence
MeSH Terms: conditions — Colitis, Ulcerative; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 5-ASA: Patient's treated with oral 5-ASA

SUMMARY:
The objectives of this study are to investigate how oral 5-ASA drugs have been used in the condition without symptoms such as abdominal pain or diarrhea/bloody stool (remission stage), or in the transition from the condition with symptoms such as abdominal pain or diarrhea/bloody stool (active stage) to the remission stage in ulcerative colitis and to study how many patients will be able to maintain the remission stage during the observation period and how many times the patients will experience the active stage (relapse), as well as how symptoms will change during the observation period to discover better treatment plans.

DETAILED DESCRIPTION:
Period: 2012-2014 Observation Time: 0, 26week, 52week

Matters investigated:

1. pUCDAI scores(Stool frequency, Bloody stool, Physician's global assessment)
2. Medication adherence (VAS scale)
3. Remission, Relapse
4. Age, gender, body height, body weight, date of diagnosis, extension of inflammation, classification by clinical course, smoking, alcohol, work, disease complication, duration of remission maintained to enrollment(remission patient)

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Adult patients who have been diagnosed with mild to moderate active ulcerative colitis or ulcerative colitis in the remission stage according to the diagnostic criteria for ulcerative colitis (draft revised on February 13, 2010)
3. Patients who have been treated with remission induction therapy or remission maintenance therapy with oral 5-ASA drugs (Pentasa® tablets 250 mg, Pentasa® tablets 500 mg, Asacol® tablets 400 mg and Salazopyrin® tablets 500 mg as well as drugs that have been proved equivalent to these drugs)
4. Patients who have received adequate information regarding this study and understood thoroughly, and then voluntarily submitted written consent forms upon participation in this study

Exclusion Criteria:

1. Patients with severe active ulcerative / fulminant ulcerative colitis according to the diagnostic criteria for ulcerative colitis (draft revised on February 13, 2012)
2. Patients who have received total / subtotal colectomy
3. Patients who have been complicated with malignant tumor
4. Patients who are pregnant or possibly pregnant
5. Other patients whom investigators and subinvestigators considered inappropriate to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University, Main hospital, General Hospital, General Practitioner
Sampling Method: Probability Sample
Enrollment: 5704 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cumulative non-relapse rate | 52 weeks

SECONDARY OUTCOMES:
Number of relapses | 52 weeks
The pUCDAI scores and the scores that constitute these pUCDAI scores at each assessment period | 0, 26 weeks, 52 weeks
Medication adherence:Measured by patient response to visual analog scale | 0, 26 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soji Omuro, Mr., Study Chair — Kyorin Pharmaceutical Co.,Ltd
Locations (1):
- Tokyo Medical and Dental University, Bunkyo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Nagahori M, Kochi S, Hanai H, Yamamoto T, Nakamura S, Omuro S, Watanabe M, Hibi T; OPTIMUM Study Group. Real life results in using 5-ASA for maintaining mild to moderate UC patients in Japan, a multi-center study, OPTIMUM Study. BMC Gastroenterol. 2017 Apr 4;17(1):47. doi: 10.1186/s12876-017-0604-y. PMID 28390410